CLINICAL TRIAL: NCT06860178
Title: Integrating Malaria Vaccine With Seasonal Malaria Chemoprevention in West Africa
Acronym: IMVACS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: R-Evolution Worldwide (Other); CNRST Burkina Faso (Unknown); USTTB Mali (Unknown); Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IMVACS
Record Dates: First submitted 2025-01-20; First posted 2025-03-05 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Malaria Vaccine
Keywords: malaria; CPS; pediatric; vaccine; R21
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Children aged 5-36 months will receive R21 via routine EPI vaccination (Year round in Burkina faso, or prior to the malaria season and SMC delivery in Mali)
- Integrated SMC Vaccination (Other): Children aged 3-59 months will receive 3-dose primary series aligned with SMC distribution in an annual campaign
  Interventions: Other: Annual campaign of the 3-dose primary series vaccine R21/Matrix-M aligned with SMC distribution in children aged 3-59 months

INTERVENTIONS:
Other: Annual campaign of the 3-dose primary series vaccine R21/Matrix-M aligned with SMC distribution in children aged 3-59 months — in the intenvention arm, the children will get the vaccine R21 Matrix M together with the CPS
  Arms: Integrated SMC Vaccination

SUMMARY:
This is a multi-site, multi-disciplinary, Phase-4 two-arm cluster-randomised non-inferiority trial in Burkina Faso and Mali to evaluate the eﬀectiveness and real-life impact of a novel integrated delivery strategy of the R21 malaria vaccine alongside SMC among children in areas with highly seasonal malaria transmission. In this study, a cluster is defined as the catchment area of a health centre. Clusters will be randomised to receive either year-round age-based routine EPI vaccination for children aged 5-36 months ("Routine EPI Vaccination") in Burkina Faso or an annual campaign of the 3-dose primary series in children aged 5-36 months prior to the malaria season and SMC delivery (''Routine Pre-SMC vaccination'') in Mali versus an annual campaign of the 3-dose primary series aligned with SMC distribution in children aged 3-59 months ("Integrated SMC Vaccination") in each country. Eﬀectiveness will be assessed in terms of clinical malaria, vaccine coverage, acceptability, feasibility, and cost-eﬀectiveness.

Malaria incidence will be determined using routine surveillance activities for clinical malaria detection and reporting in each country. Cross-sectional surveys will be conducted to determine the prevalence of parasitaemia in the communities. In addition, the acceptability, feasibility, coverage and cost-effectiveness of the different delivery systems of R21/Matrix-M will be assessed.

ELIGIBILITY:
Inclusion criteria:

Control arms :

* Children aged 5-36 months in Burkina Faso and Mali at the time of first study vaccination;
* Resident in the catchment area of a health centre assigned to the control arm;
* Willingness to comply with the study procedures;
* Written informed consent from Parent/Guardian.

Intervention arms :

* Children aged 3-59 months at the time of first study vaccination;
* Resident in the catchment area of a health centre assigned to the intervention arm;
* Willingness to comply with the study procedures;
* Written informed consent from Parent/Guardian.

Exclusion Criteria:

1. History of allergic disease or reactions likely to be exacerbated by any component of the Vaccines;
2. Any history of anaphylaxis in relation to vaccination;
3. Known chronic illness;
4. Any other significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial;
5. History of vaccination with another malaria vaccine. -

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40000 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Malaria Incidence on 5-36 months at 12 months | from enrollment to 12 months
  Malaria incidence among children aged 5-36 months over 12 months post first dose using routine surveillance activities for clinical malaria detection and reporting

SECONDARY OUTCOMES:
Malaria incidence among children aged 5-36 months over 24 and 36 months | From enrollment to 2 years after booster
  Malaria incidence among children aged 5-36 months over 24 and 36 months post first dose using routine surveillance activities for clinical malaria detection and reporting;
Malaria incidence among children aged 3-59 months over 24 and 36 months | From enrollment to 2 years after booster
  Malaria incidence among children aged 3-59 months over 24 and 36 months post first dose using routine surveillance activities for clinical malaria detection and reporting
Malaria prevalence at peak transmission | From enrollment to 2 years after booster dose
  Malaria prevalence at peak transmission in November after SMC campaigns in 2025 and 2026
Vaccine coverage | From enrollment to months 24
  Pourcentage of children who has received 3 or 4 doses at 24 months post 1st vaccination
Occurrence of adverse events (AEs) and serious adverse events (SAEs) following R21/Matrix-M vaccination; | From enrollment to months 4
  Occurrence of adverse events (AEs) and serious adverse events (SAEs) following R21/Matrix-M vaccination
Acceptability | From 12 months after study start to 36 months
  Qualitative interviews and FGDs among policy makers, health managers, health providers and caregivers
Stakeholder perceptions of the feasibility on the vaccine delivery strategy in each group | From enrollment to months 36
  Acceptability and feasibility studies will use qualitative longitudinal study (QLS) research methods. We will apply an ecological framework approach with emphasis on the interplay and inter-dependency between individual, interpersonal, organizational, and policy levels. Qualitative data will be collected through ethnographic immersion, in-depth interviews, group interviews and focus group discussions. No quantitative measurements will be made.
Contextual and behavioural factors impeding or facilitating R21/Matrix-M vaccine uptake | From enrollment to months 24
  Interviews and FGD - will be explained in a parallel protocol
Stakeholders and caregivers perceptions of the factors that enhance and/or constrain the succesful co,pletion of four doses of R21 and the key drivers of vaccination coverage | From enrollment to months 24 and 36
  The study will cover a full, two-year R21/Matrix-M delivery cycle with data collection at two time points in each arm: soon after the primary series is delivered, and soon after the booster dose is provided a year later. This longitudinal approach will enable us to explore and chart dynamic processes as they occur, barriers and facilitators, and acceptability over time. It is inherently suitable for studying R21/Matrix-M introduction, requiring prolonged and repeated involvement by patients and providers. This approach is also necessary to explore the drivers of vaccine hesitancy which is not a static state; vaccine decision-making changes over time as caregivers experience different influences and nudges along the way. Qualitative data will be collected through ethnographic immersion, in-depth interviews, group interviews and focus group discussions to explore factors in the service delivery, household, and broader social environments that will lead to R21 adoption and adherence. A
Incremental costs (per child vaccinated) and cost-effectiveness (per malaria case and separately, per DALY averted) of each vaccination strategy, calculated from a societal perspective | From enrollment to months 36
  Costs associated with the different vaccination strategies will be estimated by collecting data on direct and indirect costs to health systems and opportunity costs to vaccinees and their caregivers (beneficiaries). Beneficiary costs will be collected during household surveys, via case report forms developed to collect data on direct costs (transport, food, medication) and indirect costs (time and income loss) incurred by their household related to each intervention arm. Provider costs will be collected using custom built spreadsheets structured to comprehensively capture the resources used for all intervention delivery related activities (excluding research activities) by cost category (person time, equipment, consumables including vaccines, storage, transport, overheads and other costs) by arm. Malaria incidence estimates (primary clinical outcome) will be used to calculate malaria cases and DALYs averted by arm, adjusted for intervention coverage (using the coverage survey data).

CONTACTS AND LOCATIONS:
Locations (2):
- Institut de Recherche en Sciences de la Santé, Direction Régionale du Centre-Ouest, Ouagadougou, Burkina Faso
- University of Sciences Techniques and Technologies of Bamako, Bamako, Mali

IPD SHARING:
Plan to Share IPD: Undecided